CLINICAL TRIAL: NCT05213416
Title: VALIDITY AND RELIABILITY OF THE BETY-BIOPSYCHOSOCIAL QUESTIONNAIRE (BETY-BQ) IN PARTİCİPANTS RECEIVING RADIOTHERAPY
Brief Title: BETY-BIOPSYCHOSOCIAL QUESTIONNAIRE IN PARTİCİPANTS RECEIVING RADIOTHERAPY
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Umut Bahçacı, Principal investigator, Hacettepe University
Other Study IDs: BETY-BQ
Record Dates: First submitted 2022-01-19; First posted 2022-01-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Questionnaire; Radiotherapy
Keywords: Reliability and Validity; Biopsychosocial Models; Questionnaire; Radiotherapy; Quality of Life; Conservative Treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the validity and reliability of BETY-BQ as a biopsychosocial assessment tool in individuals receiving radiotherapy.

DETAILED DESCRIPTION:
It is known that psycho-physiological processes affect the results of medical treatment in chronic diseases [1]. In oncological rehabilitation, the psychological, social and functional problems of individuals with cancer are considered together, and goals of the treatment are determined based on this [2]. Biopsychosocial being of human is the main reason for this approach. BETY-Biopsychosocial Questionnaire (BETY-BQ) originates from the Cognitive Exercise Therapy Approach (CETA) which is an innovative exercise approach that targets a holistic treatment techniques in accordance with the biopsychosocial model [3]. This approach contains concepts including function-oriented trunk stabilization exercises, pain management, mood management (dance therapy-authentic movement), sexual knowledge management which are combined with each other. It was first used in patients with ankylosing spondylitis and was observed that besides its positive effects on disease activity, and also provided positive changes in anti-inflammatory parameters [4]. CETA has taken its place in the literature as a biopsychosocial exercise model that can be applied safely in individuals with Multiple Sclerosis [5]. Patients with rheumatism, who have participated in CETA training since 2004, described their recovery characteristics in 2013. The questionary was finalized in 2017 by applying these feedbacks to repetitive statistics and rheumatic patients who did not participate in the group [6]. Validity and reliability studies of the developed scale were conducted in individuals diagnosed with Fibromyalgia, Rheumatoid Arthritis, Osteoarthritis, and individuals with chronic neck and chronic low back pain [3, 7].

Radiotherapy reduces the recurrence rate and provides disease control in patients with cancer [8, 9] However, studies have shown that individuals receiving radiotherapy may experience treatment-related problems such as pain, limitation of movement, and even fractures [10-12]. Cognitive changes such as learning and memory, attention to the painful area, which develop with the influenced limbic system, increase the avoidance of movements. Herewith, the developing muscle spasm, pain and negative mood which results in vicious circle, can be experienced that leads to limitation of movement. Therefore, physical and psychosocial factors are also associated with musculoskeletal disorders [13]. Determining the biopsychosocial status of individuals receiving radiotherapy should be considered when evaluating the effectiveness of treatment. However, when the literature in this field is examined, it is clear that there is a need for biopsychosocial assessment tools.

In the line with this information, the aim of this study is to investigate the validity and reliability of BETY-BQ as a biopsychosocial assessment tool in individuals receiving radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with cancer
* Receiving radiotherapy from cancer treatments
* Cancer stage between 1-3
* Being between the ages of 18-70
* Having a Mini Mental Test Score of 24 and above

Exclusion Criteria:

* Not being able to read and/or understand the questionaries
* Not being willing to participate in the study
* Having a neurological disease which affects the cognition
* History of orthopaedic surgery in the last three years
* Presence of psychiatric diagnosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving radiotherapy
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire (BETY-BQ | 1 week
  It is used to evaluate the biopsychosocial process associated with the disease. A 5-point Likert system is used to score this scale. Each question is scored as "0= never, 1=yes rarely, 2=yes sometimes, 3=yes often 4=yes always" and gives a total score over 30 items. A high score means a low biopsychosocial level

SECONDARY OUTCOMES:
Quality of Life Scale Short Form-36 (SF-36) | 1 week
  It is one of the frequently used scales to measure quality of life. It evaluates 8 different categories such as general health perception, physical function, social function, pain, mental health, role difficulty due to physical reasons, role difficulty due to emotional reasons, and vitality with a total of 36 sub-items. Items are scored as '0 = worst health condition 100 = best health state'. Each subcategory is scored between 0 and 100 points, with a high score indicating good health.
Functional Assessment of Cancer Therapy-General (FACT-G) | 1 week
  It is used to evaluate the multifaceted quality of life in cancer patients; It is a general 27-item scale in which patients evaluate their own condition. There are 4 sub-scales in the questionnaire that evaluate physical, social, emotional and functional status. Participants will be asked how appropriate a particular statement was to them in the past 7 days on a 5-point scale as '0: never; 1: a little, 2: a little; 3: quite; 4: too much'. High scores indicate a high quality of life, and low scores indicate a decreased quality of life
Hospital Anxiety and Depression Scale (HADS) | 1 week
  It is a scale consisting of 14 questions which 7 of these questions assess anxiety and 7 assess depression. Likert type measurement is used to evaluate this scale. The cut-off score for the anxiety subscale is 10/11 and for the depression subscale is 7/8. Accordingly, those who score above these scores are considered at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Songül Atasavun Uysal, Prof., Study Director — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara
  - Florence Nightingale Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kline Leidy N, Ozbolt JG, Swain MA. Psychophysiological processes of stress in chronic physical illness: a theoretical perspective. J Adv Nurs. 1990 Apr;15(4):478-86. doi: 10.1111/j.1365-2648.1990.tb01843.x. PMID 2341695
- [Background] Rick O, Dauelsberg T, Kalusche-Bontemps EM. Oncological Rehabilitation. Oncol Res Treat. 2017;40(12):772-777. doi: 10.1159/000481709. Epub 2017 Nov 29. PMID 29183040
- [Background] Oflaz, F.B., Bilişsel Egzersiz Terapi Yaklaşımı Ölçeği'nin Romatoid Artrit Tanısı Alan Bireylerde Geçerliği, Güvenirliği Ve Duyarlılığının Belirlenmesi. 2018, Sağlık Bilimleri Enstitüsü.
- [Background] Kisacik P, Unal E, Akman U, Yapali G, Karabulut E, Akdogan A. Investigating the effects of a multidimensional exercise program on symptoms and antiinflammatory status in female patients with ankylosing spondylitis. Complement Ther Clin Pract. 2016 Feb;22:38-43. doi: 10.1016/j.ctcp.2015.11.002. Epub 2015 Dec 2. PMID 26850804
- [Background] Küçüktepe, İ., et al., Multiple sklerozlu bireylerde Bilişsel Egzersiz Terapi Yaklaşımı'nın yorgunluk ve denge üzerine etkileri. 2018. 5(2): p. 74-81.
- [Background] Edibe, Ü., et al., Romatizmalı hastalar için bir yaşam kalitesi ölçeğinin geliştirilmesi: madde havuzunun oluşturulması. Journal of Exercise Therapy and Rehabilitation 2017. 4(2): p. 67-75.
- [Background] ZAHİD, M., Bilişsel Egzersiz Terapi Yaklaşımı Ölçeği'nin Fibromiyalji Tanısı Alan Bireylerde Geçerliği, Güvenirliği ve Duyarlılığının Belirlenmesi. 2018, Sağlık Bilimleri Enstitüsü
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Citrin DE. Recent Developments in Radiotherapy. N Engl J Med. 2017 Sep 14;377(11):1065-1075. doi: 10.1056/NEJMra1608986. No abstract available. PMID 28902591
- [Background] Vallejo Bernad C, Casamayor Franco MDC, Perez-Tierra Ruiz JV, Martinez Lahoz Y, Carrasquer Puyal A, Pallares Segura JL, Sanchez Marin JP, Barra Pardos MV. Breast-conserving surgery in breast cancer and intraoperative radiotherapy. Can we predict the fibrosis? Cir Esp (Engl Ed). 2019 Nov;97(9):517-522. doi: 10.1016/j.ciresp.2019.05.012. Epub 2019 Jul 15. English, Spanish. PMID 31320114
- [Background] Mavrogenis AF, Papagelopoulos PJ, Romantini M, Guerra G, Ruggieri P. Side effects of radiation in musculoskeletal oncology. J Long Term Eff Med Implants. 2009;19(4):287-304. doi: 10.1615/jlongtermeffmedimplants.v19.i4.60. PMID 21083535
- [Background] Liljegren G, Holmberg L. Arm morbidity after sector resection and axillary dissection with or without postoperative radiotherapy in breast cancer stage I. Results from a randomised trial. Uppsala-Orebro Breast Cancer Study Group. Eur J Cancer. 1997 Feb;33(2):193-9. doi: 10.1016/s0959-8049(96)00375-9. PMID 9135487
- [Background] Skov T, Borg V, Orhede E. Psychosocial and physical risk factors for musculoskeletal disorders of the neck, shoulders, and lower back in salespeople. Occup Environ Med. 1996 May;53(5):351-6. doi: 10.1136/oem.53.5.351. PMID 8673184
- [Background] Koçyiğit, H., Ö. Aydemir, and G.J.R.h.o.b.g.h.i.ç.İ.v.T.D. Fişek, Kısa Form-36'nın (KF-36) Türkçe için güvenilirliği ve geçerliliği. 1999. 12: p. 102-106.
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Aydemir, O.J.T.P.D., Hastane anksiyete ve depresyon olcegi Turkce formunun gecerlilik ve guvenilirligi. 1997. 8: p. 187-280.